CLINICAL TRIAL: NCT00563849
Title: An Open-Label, Multi-Center Study to Evaluation of Leflunomide Plus Methotexate for the Treatment of Rheumatoid Arthritis in DMARDs:(Disease-Modifying Antirheumatic Drug) na¿ve or Restart (Skip DMARDs More Than 4 Weeks) Subjects.
Brief Title: Leflunomide + Methotrexate in Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HWA486_4021
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Leflunomide — concomitantly leflunomide (no loading dose, 10 mg/day) and methotrexate (starting at 7.5 mg/week and titrating up to 15 mg/week) for 20 weeks.
  Other Names: ARAVA®

SUMMARY:
To determine the efficacy and safety of the combination of leflunomide and methotrexate for treating active rheumatoid arthritis (RA) in an open noncomparative multicenter trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between ages of 18 and 75 years old.
* Female subjects must be of nonchildbearing potential (i.e., surgically sterile or at least 2 years postmenopausal) OR their participation is contingent upon the following:
* They are practicing a medically accepted contraceptive regimen (acceptable methods must include one of the following: systemic contraceptive, oral or implanted estrogen/progestin; diaphragm with intravaginal spermicide; cervical cap; intrauterine device; or condom with intravaginal spermicide) AND
* they are demonstrated not to be pregnant (by serum pregnancy test) or breast-feeding at the time of study entry AND
* they intend to continue the contraceptive regimen and remain not pregnant throughout the study AND
* they are willing to undergo pregnancy testing (serum) at screening and (urine) monthly thereafter AND
* they are fully informed as to the risks of entering the trial and provide written consent to enter the trial; female patients not sexually active should also be adequately informed about appropriate methods of contraception AND
* they agree to not get pregnant for 24 months after discontinuation of treatment with study medication or they undergo a washout procedure with cholestyramine or charcoal.
* Male subjects must consent to practice contraception during the study. The subject needs to have clinically diagnosed rheumatoid arthritis including diagnosis of RA by ACR criteria greater than or = to 6 months prior to enrollment active disease by ACR criteria . Men wishing to father a child should consider discontinuing use of study drug and taking cholestyramine 8 gm 3 times daily for 11 days. In addition, males should consider discontinuation of methotrexate treatment and waiting an additional three months.
* Active disease by ACR criteria despite methotrexate therapy for three of the following four criteria:
* greater than or = to 9 tender joints
* greater than or = to 6 swollen joints
* greater than or = to 45 minutes of morning stiffness
* ESR greater than or = to 28mm/hr

  * Subject must remain on unchanged doses of NSAIDs for at least 4 weeks prior to study drug administration and throughout the timecourse of the study.
  * Concomitant therapy will be permitted with corticosteroids at a dose of less than or = to 10 mg prednisone daily (or the steroid equivalent administered orally), provided the dose has been stable for at least 4 weeks prior to the study drug administration; dose must remain constant throughout the timecourse of the study.
  * Subjects must not receive intramuscular, intra-articular or intravenous corticosteroids within 4 weeks prior to initiating study participation or during the study.
  * Subjects must be able and willing to comply with the terms of this protocol. Informed consent must be obtained for all subjects before enrollment in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2003-05; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
The primary end point was a 20% improvement in the American College of Rheumatology criteria (ACR 20) at 20 weeks | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Choe Seong Choon, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Pusan, South Korea